CLINICAL TRIAL: NCT05651464
Title: Impact of Prophylactic Antibiotics on Bloodstream Infections After Liberation From Extracorporeal Membrane Oxygenation
Acronym: IPANEMA-ECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Philipp Lepper, Deputy Director, Universität des Saarlandes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PL002
Record Dates: First submitted 2022-11-25; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Prophylactic antibiotic treatment (Active Comparator): Application of 15-20 mg per kgKG Vancomycine I.V. prior to ECMO liberation
  Interventions: Drug: Vancomycine
- Control Arm: No prophylactic antibiotic treatment (No Intervention): Control group - no intervention.

INTERVENTIONS:
Drug: Vancomycine — Application of 15-20 mg per kgKG Vancomycine I.V. prior to ECMO liberation
  Arms: Intervention: Prophylactic antibiotic treatment

SUMMARY:
The goal of this prospective interventional study is to evaluate the impact of antibiotic prophylaxis on bloodstream infections after liberation of extracorporeal membrane oxygenation therapy. The main questions aims to answer are:

• does application of vancomycine prior to ECMO liberation have an impact of bloodstream infections?

Participants will get 1 dose of vancomycine I.V. (15-20 mg per kgKG) prior to liberation of ECMO.

Researchers will compare this interventional group to a group without antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients older than 18 years
* ECMO-Therapy

Exclusion Criteria:

* patients younger than 18 years
* fever >38,5°C
* pregnancy
* antibiotic treatment with Vancomycine, Linezolid, Daptomycin or Tygacil on the day of liberation
* prior adverse events after application of Vancomycine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth of pathogens in blood culture | taken 72 hours after liberation of extracorporeal membrane oxygenation therapy
  Detection of pathogens / blood stream infection
Growth of pathogens in blood culture | taken directly before removal of extracorporeal membrane oxygenation therapy
  Detection of pathogens / blood stream infection

SECONDARY OUTCOMES:
Growth of pathogens on cannula tip | on the day of liberation, cannula tip will be send to institute of microbiology directly after liberation from ECMO
  Detection of growth of pathogens on cannulas
laboratory parameters | 6.00 am on the day of liberation of extracorporeal membrane oxygenation therapy
  leukocytes, procalcitonin, C-reactive protein
laboratory parameters | 24 hours after liberation of extracorporeal membrane oxygenation therapy
  leukocytes, procalcitonin, C-reactive protein
laboratory parameters | 48 hours after liberation of extracorporeal membrane oxygenation therapy
  leukocytes, procalcitonin, C-reactive protein
laboratory parameters | 72 hours after liberation of extracorporeal membrane oxygenation therapy
  leukocytes, procalcitonin, C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Philipp M Lepper, MD, Principal Investigator — Saarland University Medical Center
Locations (1):
- University Hospital of Saarland, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No